CLINICAL TRIAL: NCT01784055
Title: Post-Market Surveillance Registry for the NeoChord DS1000
Brief Title: NeoChord TACT Post-Market Surveillance Registry
Status: Completed | Type: Observational
Sponsor: NeoChord (Industry)
Responsible Party: Sponsor
Other Study IDs: 800001-001
Record Dates: First submitted 2013-01-31; First posted 2013-02-05 (Estimated); Results first posted 2018-04-02 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2017-08

CONDITIONS: Mitral Valve Insufficiency; Heart Valve Diseases; Heart Diseases; Cardiovascular Diseases
Keywords: NeoChord; DS1000; Mitral Valve; Mitral Valve Regurgitation; MR; Mitral Valve Repair; Mitral Valve Prolapse; Artificial Chordae
MeSH Terms: conditions — Mitral Valve Insufficiency; Heart Valve Diseases; Heart Diseases; Cardiovascular Diseases; Mitral Valve Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

SUMMARY:
To monitor the long-term performance of the CE Marked NeoChord Artificial Chordae Delivery System

ELIGIBILITY:
Inclusion Criteria:

* Grade 3+ or 4+ mitral valve regurgitation

Exclusion Criteria:

* Heavily calcified valves
* Valvular retraction with severely reduced mobility
* Active bacterial endocarditis
* Complex mechanism of MR (leaflet perforation, etc.)
* Significant tethering of leaflets
* Inflammatory valve disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Grade 3+ or 4+ mitral valve regurgitation who are candidates for surgical mitral valve repair or replacement
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2013-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Seeberger, MD, Study Chair — Leipzig University
Locations (7):
- Bordeaux Heart University Hospital (CHU), Bordeaux, France
- Germany (3):
  - Herzzentrum Dresden, Dresden
  - Asklepios Hospital St. Georg, Hamburg
  - University Medical Center Hamburg, Hamburg
- University of Padova Medical School, Padua, Italy
- Vilniaus Universiteto ligonines Santariskiu, Vilnius, Lithuania
- Universitätsspital Basel, Basel, Switzerland

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall: All Subjects
Period: Overall Study
Arm/Group | Overall
Started | 126
Completed | 100
Not Completed | 26

BASELINE CHARACTERISTICS:
Arm/Group | Overall
Number analyzed (Participants) | 126
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One patient did not have baseline information reported
  years
    number analyzed (Participants) | 125
    (all) | 66 (14)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One patient did not have baseline information reported
  Participants
    number analyzed (Participants) | 125
    Female | 34
    Male | 91
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Procedure Success
Description: To describe the rate of subjects with at least one neochord placed using the DS1000 System AND a reduction in mitral regurgitation ≤ 2+ at the time of the procedure
Time Frame: The patient will be evaluated from the procedure through the hospital discharge. Approximately 1 day.
Measure: Count of Participants; unit: Participants
Groups:
- Overall: All patients
Arm/Group | Overall
Number analyzed (Participants) | 126
Participants
  >1 neochord placed and MR</= 2+ | 121
  No neochords placed or MR>/=3+ | 5

ADVERSE EVENTS:
Time Frame: Index procedure though 1-year follow-up visit
Arm/Group | Overall
All-Cause Mortality (participants affected / at risk) | 7/126
Serious Adverse Events (participants affected / at risk) | 37/126
Other Adverse Events (participants affected / at risk) | 9/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall (N=126)
Regurgitation (Cardiac disorders) | 2 (2)
Dyspnea (General disorders) | 2 (3)
Hepatic complication (Hepatobiliary disorders) | 1 (1)
Infection (Infections and infestations) | 3 (3)
Procedural complication (Injury, poisoning and procedural complications) | 6 (6)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neurological complication (Nervous system disorders) | 3 (3)
Renal dysfunction (Renal and urinary disorders) | 4 (4)
Respiratory complication (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Valve intervention (Surgical and medical procedures) | 13 (14)
Peripheral vascular complication (Vascular disorders) | 2 (2)
Other cardiac complication (Cardiac disorders) | 15 (19)
Other non-cardiovascular complication (General disorders) | 2 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall (N=126)
Regurgitation (Cardiac disorders) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No